CLINICAL TRIAL: NCT02028910
Title: Efficacy of Ondansetron on Vomiting Due to Acute Gastroenteritis in Pediatric During Winter
Acronym: Ondangapi
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P110105; 2011-004372- 11 (Other: N° EudraCT : 2011-004372- 11)
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2012-10

CONDITIONS: Vomiting; Gastroenteritis
Keywords: gastroenteritis; pediatrics; vomiting
MeSH Terms: conditions — Vomiting; Gastroenteritis | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ondansetron (Experimental): The treatments in the form of cases numbered 1 vial of 50 ml of ondansetron 0.8 mg / ml oral solution + 5 ml syringe for oral administration.
  No special storage conditions ondansetron syrup.The treatment is administered orally as a single dose of 2.5 ml = 2 mg per 5 kg weight of the child, not to exceed a maximum dose of 10mg. A second outlet, at the same dose, is restored if the child vomits within 15 minutes after the first administration.
  Interventions: Drug: Ondansetron
- placebo (Placebo Comparator): The treatments in the form of cases numbered 1 vial of 50 ml of placebo 0.8 mg / ml oral solution + 5 ml syringe for oral administration.
  No special storage conditions placebo syrup.The treatment is administered orally as a single dose of 2.5 ml = 2 mg per 5 kg weight of the child, not to exceed a maximum dose of 10mg. A second outlet, at the same dose, is restored if the child vomits within 15 minutes after the first administration.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — The treatment is administered orally in a single dose of 2.5 ml = 2 mg per 5 kg weight of the child, not to exceed the maximum dose of 10mg. A second dose, the same dose is given back if the child vomits within 15 minutes after the first administration.
  The bottle contains at least 2 doses of up to 10 mg for a second dose can be given back in case of vomiting within 15 minutes after the first dose in children weighing more than 25 kg.
  The dosage should be adjusted according to the weight of the child
  Other Names: Ondansetron hydrochloride dihydrate

SUMMARY:
Acute gastroenteritis is a common disease especially in children. With bronchiolitis and influenza, she participated widely in weight of winter epidemics that causes problems every year our health care system, particularly in the pediatric emergency and inpatient since they are the second leading cause of hospitalization in children. The main symptoms of viral acute gastroenteritis are diarrhea and vomiting which exposes children to the risk of sometimes severe dehydration, the most common cause of hospitalization. There is no specific treatment for these infections. At most, there is a vaccine against severe rotavirus diarrhea (Rotarix ® and RotaTeq ®), but does not yet official recommendations to use in France. The treatment of acute gastroenteritis virus is symptomatic and is generally based on the use of oral rehydration solutions (ORS) whose administration is limited by the frequent presence of vomiting. Until now, no treatment has demonstrated its effectiveness on vomiting due to acute gastroenteritis virus in children. Conventional anti-emetics, widely prescribed, are ineffective in practice, very few studies in this indication and encumbered side effects. Several drugs have long been used in children to fight against severe vomiting associated with the administration of anti-cancer chemotherapy, such as granisetron (Kytril ®) and ondansetron (Zofren ®). The mechanism of action of these molecules is well known. They act both on the enteric nervous system by blocking serotonin receptors. Several placebo-controlled trials suggest that ondansetron is effective in reducing the number of vomiting in children emergency consultant for acute gastroenteritis. However, the method used in these tests and the number of children enrolled has not yet demonstrated the efficacy of ondansetron on the number of admissions, the number of emergency and return the cost / benefit ratio of this treatment. In addition, several studies reported the occurrence of watery stools more frequently in children treated with the placebo group.

Evidence that ondansetron is well tolerated and effective for reducing the severity of vomiting during acute gastroenteritis pediatrics winter could support the use of this treatment in routine pediatric emergencies.

This study is a clinical trial, multicenter, controlled versus placebo whose main objective is to evaluate the efficacy of ondansetron to decrease the intensity of vomiting in children with acute gastroenteritis during winter emergencies Upon arrival to the emergency room after signing. Consent, an ECG is performed in eligible patients. Children meet all the criteria for inclusion and non-inclusion receive, at random, one of two treatments: ondansetron (active) or placebo. The study does not alter the usual care of the child to the emergency room. After passing emergency, patients will be followed in the study for 8 days, through a phone call home to J3 and J7. The total duration of patient participation in the study is 8 days, including 4 hours emergencies (usual transit time to emergencies).

DETAILED DESCRIPTION:
Acute gastroenteritis is a common disease especially in children. With bronchiolitis and influenza, she participated widely in weight of winter epidemics that causes problems every year our health care system, particularly in the pediatric emergency and inpatient since they are the second leading cause of hospitalization in children. The main symptoms of viral acute gastroenteritis are diarrhea and vomiting which exposes children to the risk of sometimes severe dehydration, the most common cause of hospitalization. There is no specific treatment for these infections. At most, there is a vaccine against severe rotavirus diarrhea (Rotarix ® and RotaTeq ®), but does not yet official recommendations to use in France. The treatment of acute gastroenteritis virus is symptomatic and is generally based on the use of oral rehydration solutions (ORS) whose administration is limited by the frequent presence of vomiting. Until now, no treatment has demonstrated its effectiveness on vomiting due to acute gastroenteritis virus in children. Conventional anti-emetics, widely prescribed, are ineffective in practice, very few studies in this indication and encumbered side effects. Several drugs have long been used in children to fight against severe vomiting associated with the administration of anti-cancer chemotherapy, such as granisetron (Kytril ®) and ondansetron (Zofren ®). The mechanism of action of these molecules is well known. They act both on the enteric nervous system by blocking serotonin receptors. Several placebo-controlled trials suggest that ondansetron is effective in reducing the number of vomiting in children emergency consultant for acute gastroenteritis. However, the method used in these tests and the number of children enrolled has not yet demonstrated the efficacy of ondansetron on the number of admissions, the number of emergency and return the cost / benefit ratio of this treatment. In addition, several studies reported the occurrence of watery stools more frequently in children treated with the placebo group.

Evidence that ondansetron is well tolerated and effective for reducing the severity of vomiting during acute gastroenteritis pediatrics winter could support the use of this treatment in routine pediatric emergencies.

This study is a clinical trial, multicenter, controlled versus placebo whose main objective is to evaluate the efficacy of ondansetron to decrease the intensity of vomiting in children with acute gastroenteritis during winter emergencies Upon arrival to the emergency room after signing. Consent, an ECG is performed in eligible patients. Children meet all the criteria for inclusion and non-inclusion receive, at random, one of two treatments: ondansetron (active) or placebo. The study does not alter the usual care of the child to the emergency room. After passing emergency, patients will be followed in the study for 8 days, through a phone call home to J3 and J7. The total duration of patient participation in the study is 8 days, including 4 hours emergencies (usual transit time to emergencies).

Outside the study drug administration, it will be in the framework of the research:

* An electrocardiogram inclusion
* A stool specimen
* A fill two questionnaires, one of which during the passage of emergency and the other during two phone calls within 7 days after the departure of emergencies.

This will be done in addition to the balance necessary to support the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 months and ≤ 15 years
* Children who had more than 3 non bilious vomiting and bloodless within 12 hours before emergency department visit
* Children whose parents agree to be contacted by phone
* Completion of a medical examination (to communicate results to the patient)
* Informed consent and written / holder (s) of parental authority (s) present

Exclusion Criteria:

* Children with a congenital long QT (ECG prior to inclusion required)
* Children with and / or current symptomatic cardiovascular
* Children with a shock
* Children with a concomitant surgical pathology
* Notion of head trauma within 3 days before the emergency department visit
* Suspicion of intracranial hypertension (intracranial hypertension)
* Children who underwent surgery within 14 days before the emergency department visit
* Suspected acute can be alone responsible for vomiting, such as: discovery of diabetes, acute adrenal insufficiency, including acute neurological acute meningitis, acute respiratory illness with cough emetogenic acute otitis media, acute pyelonephritis, .. . .
* Child tracking to one of the following chronic conditions treated:

heart o

* pulmonary
* digestive (except gastroesophageal reflux)
* kidney
* hematologic (immunosuppression / SCD)
* endocrine / metabolic (diabetes, adrenal insufficiency)

  * Phenylketonuria
  * Allergy or intolerance to ondansetron or any of the ingredients of the syrup
  * Children who received treatment with an anti-emetic (Primperan ®, Motilium ®, vogalene ®) within 24 hours before emergency department visit
  * Pregnancy or breastfeeding
  * No affiliation to a social security scheme (beneficiary or assignee)
  * Family not speaking

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Success will be defined by the absence of vomiting between 15 minutes and 4 hours after administration of study treatment. | the absence of vomiting between 15 minutes and 4 hours after administration of study treatment.
  Success will be defined by the absence of vomiting between 15 minutes and 4 hours after administration of study treatment.

SECONDARY OUTCOMES:
Hospital admissions for acute gastroenteritis, intravenous infusion for rehydration, return emergency department visit, severity and duration of diarrhea and vomiting. Treatment safety will also be assessed. These criteria will be assessed within 7 days | These criteria will be assessed within 7 days after the departure of emergencies.
  Hospital admissions for acute gastroenteritis, intravenous infusion for rehydration, return emergency department visit, severity and duration of diarrhea and vomiting. Treatment safety will also be assessed.
  These criteria will be assessed within 7 days after the departure of emergencies.

CONTACTS AND LOCATIONS:
Overall Officials: Gajdos Vincent, PHD, Principal Investigator — APHP
Locations (1):
- Vincent Gajdos, Clamart, Clamart, France